CLINICAL TRIAL: NCT02383849
Title: IMPAACT P1106: Pharmacokinetic Characteristics of Antiretrovirals and Tuberculosis Medicines in Low Birth Weight Infants
Status: Completed | Type: Observational
Sponsor: International Maternal Pediatric Adolescent AIDS Clinical Trials Group (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IMPAACT P1106; 11882 (Other: DAIDS)
Record Dates: First submitted 2014-10-22; First posted 2015-03-09 (Estimated); Last update posted 2021-08-06 (Actual); Status verified 2020-03

CONDITIONS: Low-Birth-Weight Infant; Tuberculosis; HIV
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cell pellets from PK sampling once will be combined and stored for a DNA extraction, amplification, and gel electrophoresis. The genotype analysis will be completed one time per study participant. All subjects receiving INH will be genotyped for NAT2. All subjects receiving NVP will be genotyped for CYP 2B6. These genotypes will be used as covariates in the population PK analyses of NVP and INH to determine their impact on CL/F (clearance [apparent]).
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (6):
- Arm 1: Breastfeeding infants 7 to 14 days of age with birth weight less than 2500 grams born to HIV-infected mothers not receiving maintenance ARV therapy including NVP; Mother HIV-infected and TB negative; infant receiving NVP prophylaxis but not TB prophylaxis or treatment
- Arm 2: Breastfeeding infants 7 to 84 days of age with birth weight less than or equal to 4000 grams born to HIV-infected mothers not receiving maintenance ARV therapy including NVP; Mother HIV-infected with active TB disease; infant receiving NVP prophylaxis plus isoniazid (INH) but not rifampicin (RIF) for TB prophylaxis
- Arm 3: Breastfeeding infants 7 to 14 days of age with birth weight less than 2500 grams born to HIV-infected mothers not receiving maintenance ARV therapy including NVP; Mother HIV-infected with active TB disease; infant receiving NVP prophylaxis plus INH plus RIF for TB prophylaxis or treatment
- Arm 4: Breast or formula feeding infants 7 to 84 days of age with birth weight less than or equal to 4000 grams born to HIV-uninfected mothers with active TB disease; infant receiving INH alone or INH plus RIF for TB prophylaxis
- Arm 5: Breast or formula feeding infants newly diagnosed with HIV infection weighing less than or equal to 4000 grams at birth and are less than or equal to 12 weeks of age. Infants who were enrolled in Arms 1, 2 or 3 and later determined to be HIV infected are then are eligible to enroll in Arm 5 if started on an LPV/r regimen. Infants initiating treatment with LPV/r plus 2 NRTIs, and not receiving RIF (but may be receiving INH)
- Arm 6: Breast or formula feeding infants newly diagnosed with HIV infection weighing less than 2500 grams at birth and are less than or equal to 12 weeks of age. Infants who were enrolled in Arms 1, 2 or 3 and later determined to be HIV infected are then are eligible to enroll in Arm 6 if started on an LPV/r regimen. Infants initiating treatment with LPV/r plus 2 NRTIs, and receiving RIF (and may be receiving INH)

SUMMARY:
P1106 is Phase IV prospective pharmacokinetic (PK) study of low birth weight infants who are receiving or will be receiving as part of clinical care nevirapine (NVP) prophylaxis, tuberculosis (TB) prophylaxis or treatment and/or combination antiretroviral (ARV) treatment containing lopinavir/ritonavir (LPV/r). The study is designed to describe the pharmacokinetics and safety of NVP, INH, RIF, and LPV/r in these infants receiving the drug(s) as part of clinical care.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria for Arms 1 and 3 (HIV-exposed infants):

* Breastfeeding infants born to HIV-infected mothers who are receiving either no ARV therapy or ARV therapy that does not include NVP
* Age 7 to 14 days
* Birth weight less than 2500 grams
* Receiving or will be receiving prophylaxis as prescribed by clinical care provider as follows: NVP (Arm 1), NVP plus INH (Arm 2), NVP plus INH plus RIF (Arm 3)
* Parent or legal guardian able and willing to provide written informed consent. [Note to sites: modify per locally relevant language].

Inclusion Criteria for Arm 2 (HIV-exposed infants):

* Breastfeeding infants born to HIV-infected mothers who are receiving either no ARV therapy or ARV therapy that does not include NVP
* Age 7 to 84 days
* Birth weight less than or equal to 4000 grams
* Receiving or will be receiving prophylaxis as prescribed by clinical care provider as follows: NVP (Arm 1), NVP plus INH (Arm 2), NVP plus INH plus RIF (Arm 3)
* Parent or legal guardian able and willing to provide written informed consent. [Note to sites: modify per locally relevant language].

Inclusion Criteria for Arm 4 (HIV-unexposed but TB exposed infants):

* Age 7 to 84 days
* Birth weight less than or equal to 4000 grams
* Receiving prophylaxis with INH alone or INH plus RIF as prescribed by clinical care provider
* Not receiving any therapy for HIV prophylaxis or treatment
* Parent or legal guardian able and willing to provide written informed consent. [Note to sites: modify per locally relevant language].

Inclusion Criteria for Arms 5 and 6 (HIV-infected infants):

* Documentation of HIV-1 infection defined as positive HIV DNA PCR done as part of clinical care. An HIV RNA confirmatory test must be done at study entry but results may be pending at time of enrollment.
* Birth weight less than or equal to 4000 grams
* Age less than or equal to 12 weeks (defined as 84 days)
* Intention by clinical care provider to prescribe LPV/r plus 2 NRTIs and no RIF (Arm 5) or LPV/r plus 2 NRTIs plus RIF (Arm 6)
* Parent or legally acceptable representative able and willing to provide written informed consent. [Note to sites: modify per locally relevant language].

Exclusion Criteria:

Any severe congenital malformation or other medical condition incompatible with life or that would interfere with study participation or interpretation, as judged by the examining clinician.

Ages: 7 Days to 84 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Low birth weight (LBW) infants less than or equal to 2500 grams at birth who are receiving or will be receiving as part of clinical care nevirapine (NVP) prophylaxis, tuberculosis (TB) prophylaxis or treatment and/or combination antiretroviral (ARV) treatment containing lopinavir/ritonavir (LPV/r)
Sampling Method: Non-Probability Sample
Enrollment: 124 (Actual)
Dates: Start 2015-08-04 (Actual); Primary Completion 2020-02-14 (Actual); Study Completion 2020-02-14 (Actual)

PRIMARY OUTCOMES:
Clearance of NVP, INH, RIF, and LPV/r after oral dose | Week 24 of life
  Apparent clearance (CL/F) of NVP, INH, RIF, and LPV/r

SECONDARY OUTCOMES:
Primary safety endpoints | Study duration
  Number of participants with adverse events of grade 3 or 4 severity, death, or serious adverse clinical events

CONTACTS AND LOCATIONS:
Overall Officials: Mark Cotton, MD, MBChB, FCPaed, MMED, Study Chair — University of Stellenbosch; Mark H Mirochnick, MD, Study Chair — Boston Medical Center
Locations (2):
- South Africa (2):
  - Soweto IMPAACT CRS (8052), Johannesburg, Gauteng
  - Family Clinical Research Unit (FAM-CRU) CRS (8950), Cape Town, Western Cape

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 3 months following publication and available throughout period of funding of the International Maternal Pediatric Adolescent AIDS Clinical Trial (IMPAACT) Network by NIH.
Access Criteria: * With whom? Researchers who provide a methodologically sound proposal for use of the data that is approved by the IMPAACT Network.
  * For what types of analyses? To achieve aims in the proposal approved by the IMPAACT Network.
  * By what mechanism will data be made available? Researchers may submit a request for access to data using the IMPAACT "Data Request" form at: https://www.impaactnetwork.org/studies/submit-research-proposal. Researchers of approved proposals will need to sign an IMPAACT Data Use Agreement before receiving the data.

REFERENCES:
- [Derived] Bekker A, Yang J, Wang J, Cotton MF, Cababasay M, Wiesner L, Moye J, Browning R, Nakwa FL, Rabie H, Violari A, Mirochnick M, Cressey TR, Capparelli EV. Safety and Pharmacokinetics of Lopinavir/Ritonavir Oral Solution in Preterm and Term Infants Starting Before 3 Months of Age. Pediatr Infect Dis J. 2024 Apr 1;43(4):355-360. doi: 10.1097/INF.0000000000004243. Epub 2024 Jan 4. PMID 38190642